CLINICAL TRIAL: NCT02811887
Title: A Randomized, Pragmatic, Outcome-assessor-blinded Study of an SMS-message-based Lifestyle Intervention in Patients With Decompensated Liver Cirrhosis
Brief Title: SMS-based Lifestyle Intervention for Patients With Liver Cirrhosis With Previous Hepathic Encephalopathy
Acronym: SMILE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment of study participants
Sponsor: Marius Henriksen (Other)
Responsible Party: Sponsor-Investigator, Marius Henriksen, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FYS003; H-16025360 (Other: The Committees on Health Research Ethics in the Capital Region of Denmark)
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Liver Cirrhosis, Alcoholic
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): 12 weeks of supervised physical exercise followed by usual care in the outpatient liver cirrhosis rehabilitation clinic
  Interventions: Behavioral: Supervised exercise; Other: Usual Care
- SMS-messages (Experimental): 12 weeks of supervised physical exercise followed by usual care in the outpatient liver cirrhosis rehabilitation clinic + regular text messages via SMS over a 12-week period
  Interventions: Behavioral: Supervised exercise; Behavioral: SMS-messages

INTERVENTIONS:
Behavioral: Supervised exercise — A 12 week supervised and facility-based exercise training program. The program is facility based and supervised by a physiotherapist. The program runs 3 times weekly for 12 weeks. The exercise is group-based. The exercise program lasts approximately 1 hour and consists of a brief warm-up phase (bicycle ergometer at moderate intensity) followed by a circuit training program focusing on strength and endurance exercises of the large muscle groups (e.g. quadriceps).
Other: Usual Care — Participants allocated to usual care will receive instructions related to healthy living, alcohol absenteeism, and benefits of increased physical activity. The instructions will be provided by a physical therapist and/or a nurse, and will be given according to recommendations and local and national guidance. The participants are offered continued regular visits at the rehabilitation clinic, but no supervised physical exercise.
  Arms: Usual care
Behavioral: SMS-messages — Participants allocated to SMS-messages will receive the same intervention as usual care (see above) AND regular text messages via SMS over a 12-week period.
  The text messages will be unidirectional and will serve as motivational information but will not allow two-way communication with a researcher or health professional about clinical management. The messages will provide information, motivation, and support to adhere to a healthy lifestyle, alcohol absenteeism, and physical activity and will reinforce the information and instructions received at the face-to-face information (usual care).
  Arms: SMS-messages

SUMMARY:
To investigate whether simple reminders about healthy lifestyle sent via mobile phone text messages can improve the liver cirrhosis severity and prognosis (as assessed by the MELD score supported by the Child-Pugh score) among patients with liver cirrhosis that have been through a 12-week supervised and facility-based physical exercise training program and in-patient rehabilitation.

DETAILED DESCRIPTION:
Physical exercise and other interventions focused on lifestyle factors have not only the potential to increase physical functioning and capacity, but also to affect fundamental aspects of disease, increase quality of life, and may even increase survival in patients with liver cirrhosis.

Instruction and advice about a healthy lifestyle and physical activity are attractive as it limits time spent on supervised rehabilitation at an outpatient clinic. Further, self-management can be attractive to society as it can conserve health care resources. However, instructions and advice can only be effective if the patients adhere to them, and there is a need for initiatives that enhance the motivation to follow the advice and change undesirable behaviours.

Mobile phone short-message service (SMS) messages are increasingly used to deliver interventions and enhance healthy behaviour. The technology is simple, cost-effective, can be automated, and can reach any mobile phone owner. In a recent systematic review, SMS-messages have been shown effective in a broad range of healthy behaviours, which was also highlighted in a randomized trial showing positive effects of lifestyle-focused SMS-messages on cardiovascular risk factors in patients with coronary heart disease. An SMS-message-based lifestyle intervention therefore seems like a feasible and effective means of enhancing motivation to follow advice about healthy lifestyle and physical activity among patients with liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, i.e. age 18 years or above.
2. Is attending the liver cirrhosis rehabilitation clinic at Bispebjerg hospital; i.e., has alcohol-induced liver cirrhosis or hepatorenal syndrome and has at least once experienced severe decompensation in the form of hepatic encephalopathy or variceal haemorrhage.
3. Has attended at least 50% of the scheduled sessions in the 12 week run-in physical exercise program
4. Is the owner of a mobile phone capable of receiving SMS-messages
5. Has signed informed consent
6. Reads and speaks Danish

Exclusion Criteria:

1. Any condition that in the opinion of the investigator puts an otherwise eligible participant at increased risk by participation or otherwise make the person unfit for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-08; Primary Completion 2019-10 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in The Model for End-Stage Liver Disease (MELD) score | week -12, 0, 12, 24
  The MELD is a reliable measure of mortality risk in patients with end-stage liver disease. The MELD is based on a mathematical equation.
  The MELD score is calculated using the following formula:
  MELD Score = 9.57 x ln (creatinine mg/dL) + 3.78 x ln(bilirubin mg/dL) + 11.2 x ln(INR)+ 6.43

SECONDARY OUTCOMES:
10.2.1.1 Child-Pugh score | week -12, 0, 12, 24
Quality of life, SF-36v1 | week -12, 0, 12, 24
  10.2.2.1 Quality of life, SF-36v1 Short Form-36v1 is a standardised patient-reported instrument for use as a measure of health outcome and quality of life
SOKRATES questionnaire | week -12, 0, 12, 24
  SOKRATES8a is a standardised patient-reported instrument for use as a measure of readiness for change in alcohol abusers
Sickness Impact Profile (SIP) questionnaire | week -12, 0, 12, 24
  The Sickness Impact Profile (SIP) questionnaire is a 136 items generic health status measure
Six-Minute Walk Test | week -12, 0, 12, 24
  The Six-Minute Walk-Test (6MWT) assesses general physical function. The test is performed in an undisturbed hospital corridor marked every 2 meters with coloured tape on the floor; starting and turning points marked by cones. Subjects are instructed to walk as fast as they can. They are allowed to stop or rest during the test if necessary and walking aids are allowed. The distance in meters covered during the 6 minutes is the outcome of the test.
30-seconds chair stand test | week -12, 0, 12, 24
  The 30-seconds chair stand test (30-s CST) is performed in an undisturbed room with hands crossed against the chest. It is one of the most important functional evaluation clinical tests because it measures lower body strength and relates it to the most demanding daily life activities. A 30-s CST consists of standing up and sitting down from a chair as many times as possible within 30 seconds.
Muscle Power | week -12, 0, 12, 24
  The Leg Extensor Power Rig will be used to measure muscle power (force x velocity) in a non-invasive way. The participants will be in a seated position and a single explosive limb extension will accelerate a flywheel from rest. The participants will be instructed to kick the pedal as hard and fast as possible. Repeated kicks are performed, until a significant decline in power is observed. The kick with maximal power is the result of the text, and is recorded in Watts.
Standard blood sample | week -12, 0, 12, 24
  As part of the usual assessment of the patients, standard blood samples (15ml) are drawn and analysed (4 visits x 15 ml = 60 ml per participant). The analyses include: Haemoglobin (Hgb), white blood cells, Bilirubin, ALAT, ASAT, INR, platelets, CRP, creatinine, urea, sodium, potassium, alkaline phosphatase albumin, coagulations factors II VII and X.
Plasma concentrations of inflammatory markers | week -12, -6, 0
  EDTA plasma will be collected at before and after 12 weeks of supervised training intervention, and before and after a single exercise session in week 6 to analyse specific for cytokines/myokines interactions e.g. TNF alfa and IL-6.

OTHER OUTCOMES:
Continuous Reaction Time | week -12, 0, 12, 24
  Continuous Reaction Time (CRT) is a 10-minute computer-based test measuring the patient's reaction-time to a beep-sound and the patient's ability to concentrate. CRT-index below 1.9 is compatible with minimal hepatic encephalopathy .
Portosystemic Encephalopathy test | week -12, 0, 12, 24
  The Portosystemic Encephalopathy test (PSE) measures complex cognitive functions such as attention, accuracy, working speed, and visual orientation. It is a paper-and-pencil test consisting of five subtests: Digit Symbol test, Number Connection Test A, Number Connection Test B, Serial Dotting Test, and Line Tracing Test. Calculating the test score from the seconds spent on each subtest takes 5 minutes. The summed test score, the portosystemic hepatic encephalopathy score (PHES), ranges from 218 to 6, and a result below 24 is abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Christian H Dall, PhD, Study Chair — University Hospital Bispebjerg and Frederiksberg; Nanna M Jensen, PhD, Principal Investigator — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- Bispebjerg Hospital, Department of Physical and Occupational Therapy, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided